CLINICAL TRIAL: NCT05584943
Title: Kinetics of Circulating Extracellular Vesicles Over the 24-hour Dosing Interval After Low-dose Aspirin Administration in Patients at Cardiovascular Risk
Brief Title: Kinetics of cEVs Over the 24-hour Dosing Interval After Low-dose Aspirin Administration
Status: Completed | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Francesca Santilli, Associate Professor of Internal Medicine, Department of Medicine and Aging, Head of Thrombosis and Hemostasis Unit, G. d'Annunzio University
Other Study IDs: EvASA
Record Dates: First submitted 2022-10-04; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Cardiovascular Diseases; Vesicle
Keywords: circulating extracellular vesicles; aspirin
MeSH Terms: conditions — Cardiovascular Diseases; Blister

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 84 patients on ASA chronic treatment: A total of 84 patients on chronic treatment with low-dose ASA (enteric coated, Cardio aspirin 100 mg/die Bayer, Milan, Italy) once daily (o.d.) for at least 1 month
- Healthy subject: 9 healthy subjects, not on ASA treatment, as controls.

SUMMARY:
Extracellular vesicles (EVs) are small vesicles deriving from all cell types during cell activation, involved in transcellular communication, and regarded as predictors of vascular damage and of cardiovascular events. The investigators will test the hypothesis that, in patients on chronic low-dose aspirin treatment for cardiovascular prevention, aspirin may affect the release of EVs within the 24 hours interval.

ELIGIBILITY:
Inclusion Criteria:

* patients on low-dose aspirin treatment for cardiovascular prevention for at least 1 month
* arterial hypertension if well controlled with stable drug therapy
* hypercholesterolemia if well controlled with stable drug therapy

Exclusion Criteria:

* cigarette smoking insufficiency
* clinically significant hepatic insufficiency
* clinically significant renal insufficiency
* clinically significant cardiac insufficiency
* clinically significant pulmonary insufficiency
* history of malignant neoplasms (diagnosed and treated within the past 5 years)
* pregnancy or lactation
* history of malabsorption
* regular (daily) alcohol consumption
* regular (i.e., more than 3 days per week) non steroidal anti-inflammatory drug intake
* type 1 diabetes excluded by islet autoantibodies evaluation (anti-glutamic acid decarboxylase, islet cell cytoplasmic, and IA-2 antibodies), family history of type 1 diabetes, age lower than 40 years, lean phenotype, early requirement for insulin therapy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients on low-dose aspirin treatment for cardiovascular prevention (enteric coated, Cardio aspirin 100 mg/die Bayer, Milan, Italy) once daily (o.d.) for at least 1 month
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2015-09-21; Primary Completion 2017-05-09 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Kinetics of circulating extracellular vesicles after low-dose aspirin administration | 1st - 12th month
  In patients receiving low-dose aspirin for cardiovascular prevention, evaluate the potential effects of chronic aspirin treatment on circulating extracellular vesicles levels over the 24-hour interval
Aspirin response and circulating extracellular vesicles over the 24-hour | 13th - 24th month
  In patients receiving low-dose aspirin for cardiovascular prevention, evaluate the role of circulating extracellular vesicles as a potential determinant of interindividual variability in the aspirin response